CLINICAL TRIAL: NCT04629547
Title: Sleep Trial to Prevent Alzheimer's Disease
Acronym: SToP-AD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Good Ventures (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Brendan Lucey, Principal Investigator, Sleep Medicine Section Head, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202008007
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Sleep; Alzheimer Disease
Keywords: poor sleep; Amyloid-Beta; Insomnia
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid; Sleep Initiation and Maintenance Disorders | interventions — suvorexant; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Poor sleep treatment group (Experimental): 100 participants will be randomized to take suvorexant 20mg daily at h.s. for 18-24 months
  Interventions: Drug: Suvorexant 20 mg
- Poor sleep control grop (Placebo Comparator): 100 participants will be randomized to take placebo daily at h.s. for 18-24 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant 20 mg — Suvorexant 20mg will be taken nightly for 24 months.
  Other Names: Belsomra
  Arms: Poor sleep treatment group
Drug: Placebo — Placebo will be taken nightly for 24 months.
  Other Names: inactive pill; sugar pill
  Arms: Poor sleep control grop

SUMMARY:
The purpose of this study is to determine if treatment with the sleep aid suvorexant can decrease the rate of amyloid-β (Aβ) accumulation in the brain.

DETAILED DESCRIPTION:
This study will investigate if long-term treatment with suvorexant will slow amyloid-β accumulation in the brain. Amyloid-β is a protein involved in the disease process leading to Alzheimer's disease. This study will evaluate if suvorexant can decrease the amount of amyloid-beta detected by plasma pT217/T217.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Any race or ethnicity.
* Participants must be age ≥65 years and able to sign informed consent.
* Global Clinical Dementia Rating (CDR) 0.
* Willing and able to undergo study procedures.

Exclusion Criteria:

* History of reported symptoms suggestive of restless legs syndrome, narcolepsy or other central disorder of hypersomnolence, or parasomnia
* STOP-Bang score >6 for participants without PAP
* Untreated OSA with AHI ≥15 on home sleep test
* Treated sleep apnea with PAP non-compliance

  * PAP compliance is defined as >= 4 hours per night >70% of the nights
* Plasma A-beta and tau test with a plasma p-tau 217% ≤ 1.19
* Stroke.
* Chronic kidney disease defined as patients with markers of kidney damage or eGFR of < 45 ml/min/1.73m2.
* Hepatic impairment defined as AST and/or ALT > 2x upper limit of normal (normal limits AST: 11-47 IU/L, ALT: 6-53 IU/L).
* HIV/AIDS.
* History of substance abuse or alcohol abuse in the proceeding 6 months.
* Regular alcohol consumption 3 or more days a week over the last 6 months. Regular alcohol consumption is defined as having more than 2 alcoholic beverages within 3 hours of bedtime. Participants that agree to reduce alcohol consumption during the study may not be excluded.
* History of presence of any clinically significant medical condition, behavioral or psychiatric disorder, or surgical history based on medical record or participant report that could affect the safety of the participant or interfere with study assessments or in the judgement of the Principal-Investigator (PI) if participant is not a good candidate.
* Has any medical condition that, in the PI's opinion, could increase risk to the participant, limit the participant's ability to tolerate the research procedures, or interfere with the collection/analysis of the data. Potential medical conditions that will be exclusionary at the PI's discretion:

  * Cardiovascular disease requiring medication except for controlled hypertension.
  * Pulmonary disease.
  * Type I diabetes.
  * Neurologic or psychiatric disorder requiring medication.
  * Tobacco use.
  * Use of sedating medications.
  * Use of medications that interact with suvorexant (if cannot be discontinued)
  * Abnormal safety labs
* History of current suicidal ideations.
* Currently pregnant or breast-feeding.
* In the opinion of the PI, the participant should be excluded due to an abnormal physical examination.
* Must not have participated in any clinical trial involving a study drug or device within the 30-days prior to study enrollment.
* Must not participate in another drug or device study prior to the end of this study participation.

Exclusion criteria for optional lumbar punctures

-• Contraindication to lumbar puncture (anticoagulants; bleeding disorder; allergy to lidocaine or disinfectant; prior central nervous system or lower back surgery).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Amyloid-β accumulation measured by plasma pT217/T217 in participants treated with 20 mg suvorexant compared to placebo | 18-24 months
  Blood collection

SECONDARY OUTCOMES:
Change in plasma Amyloid-β compared to placebo | 18-24 months
  Blood collection
Change in CSF Amyloid-β compared to placebo | 18-24 months
  Cerebrospinal fluid collection
Change in plasma tau compared to placebo | 18-24 months
  Blood collection
Change in CSF tau compared to placebo | 18-24 months
  Cerebrospinal fluid collection
Change in plasma p-tau compared to placebo | 18-24 months
  Blood collection
Change in CSF p-tau compared to placebo | 18-24 months
  Cerebrospinal fluid collection
Change in cognitive performance compared to placebo | 18-24 months
  Measured by a cognitive composite consisting of the Digit Symbol Substitution Test, Animal Naming, Trails B and the Free and Cued Selective Reminding Test. Each test will be z-scored and then averaged together to make the composite.
Change in transcriptomics compared to placebo | 18-24 months
  blood and optional CSF collection
Change in metabolomics compared to placebo | 18-24 months
  blood and optional CSF collection
Change in proteomics compared to placebo | 18-24 months
  blood and optional CSF collection
Change in gut microbiome compared to placebo | 18-24 months
  optional stool sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Lucey, MD, Principal Investigator — Washington Univeristy School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States